CLINICAL TRIAL: NCT06213701
Title: Comparing the Healthy Minds Program With an Active Control and Waitlist Control in Depression: Pilot Study
Brief Title: Behavior, Biology and Well-Being Study
Acronym: BeWell
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Hope for Depression Research Foundation (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-0991: Pilot; Protocol Version 6/29/2023 (Other: UW Madison); A487400 (Other: UW Madison); 1U24AT011289-01 (NIH)
Record Dates: First submitted 2024-01-09; First posted 2024-01-19 (Actual); Results first posted 2025-05-02 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-04

CONDITIONS: Depression; Psychological Distress
Keywords: inflammation; microbiota; alpha diversity
MeSH Terms: conditions — Depression; Inflammation

STUDY DESIGN:
Intervention Model Description: The groups will be randomized to one of three groups in a 2:2:1 ratio.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy Minds Program (HMP) app (Experimental): Participants will receive access to the 4-week HMP Foundations module. The HMP app is a meditation-based smartphone app designed to promote and protect psychological well-being through sustainable skills training. The program is grounded in constituents of psychological well-being identified in empirical literature. HMP provides core content, with instruction administered through a curriculum of guided practices. HMP is based on research on eudaimonic well-being (e.g., environmental mastery, purpose) and brain-based skills that underlie these qualities (e.g., regulation of attention, mental flexibility). The full HMP has guided audio practices that address 4 constituents of well-being: awareness, connection, insight, and purpose. At post-treatment, participants will be given access to additional HMP content to support their continued practice.
  Interventions: Device: Healthy Minds Program
- Psychoeducation app (Active Comparator): Participants will receive access to the 4-week HMP Foundations module with guided meditation practices removed. The active control will include only the didactic content included in HMP without the guided meditation practices.
  Interventions: Other: Psychoeducation app
- Usual Care (No Intervention): Participants will receive access to HMP at the end of the study and will be encouraged to continue with their usual care.

INTERVENTIONS:
Device: Healthy Minds Program — HMP is a 4-week mobile health (mHealth) meditation training program.
  Other Names: HMP
  Arms: Healthy Minds Program (HMP) app
Other: Psychoeducation app — Psychoeducation app
  Arms: Psychoeducation app

SUMMARY:
The central aim of this pilot study is to compare markers of inflammation and gut microbial diversity with users of the Healthy Minds Program (HMP) app, an intervention designed to promote well-being. The investigators plan to conduct a randomized controlled trial (RCT) involving 300 participants comparing 4-weeks of the HMP app with an active control (Psychoeducation [HMP without meditation practice]), and a waitlist control in a sample of United States adults with elevated depression symptoms.

DETAILED DESCRIPTION:
Depression is highly prevalent and associated with extreme personal and societal costs. Meditation training reduces depression symptoms and psychological distress, but access to in-person programs is limited due to associated cost and lack of available services. Research on neurocognitive and biological mechanisms of mediation training in alleviating depression is at a preliminary stage, and an obstacle limiting research progress is over-reliance on retrospective self-report measures, which are vulnerable to a host of biases. This project will use gold-standard behavioral measures and explore novel measures of relevant neurocognitive and behavioral processes, namely pattern separation, self-referential thought, and video-based assessment of emotional well-being. Furthermore, the project will investigate effects on the gut microbiome (with fecal samples) and inflammation (with dried blood spots), which reflect biological systems hypothesized to be mechanistically related to benefits of meditation and well-being training.

Specific Aims:

* Aim 1. Determine the feasibility and acceptability of assessing inflammatory activity and gut microbiome within the context of a fully remote randomized controlled trial (RCT). Participants with elevated depression symptoms from an RCT (n = 1,100; registered to NCT05183867) comparing the Healthy Minds Program (HMP) app with an active control (HMP with didactic content only) and wait-list will be invited to provide dried blood spots (DBS) for inflammatory protein analysis and fecal samples for gut microbial analysis at baseline and 3-month follow-up. Hypotheses: It will be feasible to recruit 300 participants to provide DBS and fecal samples and 80% will provide samples at both time points (completer n = 240) with no differences in completion rates between non-Hispanic White and racial/ethnic minority participants.
* Aim 2. Characterize the association between self-reports of well-being, inflammatory activity at baseline, and microbiota diversity at baseline. Hypotheses: Well-being will correlate inversely with both protein biomarkers of inflammation (CRP, IL-6) and mRNA-derived indicators of pro-inflammatory transcriptional activity. Well-being will correlate positively with alpha diversity of the gut microbiome. These associations will not be moderated by participant race/ethnicity.
* Aim 3. Evaluate intervention effects on inflammatory activity and microbiota diversity. Hypotheses: Participants randomized to HMP or the active control will show larger reductions in inflammation vs. wait-list at 3-month follow-up and larger increases in alpha diversity of the gut microbiome vs. wait-list at 3-month follow-up. HMP will show larger reductions in inflammation vs. active control at 3-month follow-up and larger increases in alpha diversity vs. active control at 3-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Elevated PHQ-8 or PHQ-9 ≥ 5 at screening and pre-baseline interview
* Proficient in English
* Able to provide informed consent
* Have access to a smartphone that can download apps from Google Play or the Apple App Store
* For payment purposes, must be a US citizen or a permanent US resident

Exclusion Criteria:

* Regular daily meditation practice for past 6 months or regular weekly meditation practice for past 12 months
* Attended a meditation retreat or a yoga/body practice retreat with a significant meditation component

  - Previous use of Healthy Minds Program app
* Current suicidal intent and/or high self-injury risk (determined from the interview)
* Self-reported history of psychosis
* Self-reported history of mania
* Current psychopathology that interferes with study participation as assessed by interview
* Living or traveling outside the US during the whole study participation period (trips outside US after the interview phase is not an exclusion)
* Alcohol Use Disorders Identification Test (AUDIT) score ≥ 13 for women and AUDIT score ≥ 15 for men
* Drug Use Disorders Identification Test (DUDIT) score ≥ 8 for women and men

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2022-06-16 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Goldberg, PhD, Principal Investigator — UW-Madison, Center for Healthy Minds
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: FULL Behavior, Biology and Well-Being Study — https://clinicaltrials.gov/study/NCT05183867

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Started | 120 | 122 | 58
Completed | 118 | 121 | 58
Not Completed | 2 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Healthy Minds Program (HMP) App: Participants will receive access to the 4-week HMP Foundations module. The HMP app is a meditation-based smartphone app designed to promote and protect psychological well-being through sustainable skills training. The full HMP has guided audio practices that address 4 constituents of well-being: awareness, connection, insight, and purpose. At post-treatment, participants will be given access to additional HMP content to support their continued practice.
- Total: Total of all reporting groups
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care | Total
Number analyzed (Participants) | 120 | 122 | 58 | 300
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.26 (11.77) | 38.70 (11.76) | 43.57 (12.00) | 40.26 (11.90)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Man | 23 | 29 | 11 | 63
  Woman | 94 | 91 | 46 | 231
  Other | 2 | 1 | 1 | 4
  Not Provided | 1 | 1 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 90 | 98 | 38 | 226
  Racial/Ethnic Minority | 30 | 24 | 20 | 74
Region of Enrollment [Number; unit: participants]
  United States | 120 | 122 | 58 | 300

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of DBS Collection as Measured by Number of Participants Who Provide DBS
Description: Feasibility is defined as 80% of participants providing samples at both time points (completer n = 240) with no differences in completion rates between non-Hispanic White and racial/ethnic minority participants.
Time Frame: Baseline and 3 month follow-up
Measure: Count of Participants; unit: Participants
Groups:
- Non-Hispanic White: HMP App; Racial / Ethnic Minority: HMP App: Study Intervention - Participants will receive access to the 4-week HMP Foundations module.
- Non-Hispanic White: Psychoeducation App; Racial / Ethnic Minority: Psychoeducation App: Active Control - Participants will receive access to the 4-week HMP Foundations module with guided meditation practices removed. The active control will include only the didactic content included in HMP without the guided meditation practices.
- Non-Hispanic: Usual Care; Racial / Ethnic Minority: Usual Care: Usual Care: Participants will receive access to HMP at the end of the study and will be encouraged to continue with their usual care.
Arm/Group | Non-Hispanic White: HMP App | Racial / Ethnic Minority: HMP App | Non-Hispanic White: Psychoeducation App | Racial / Ethnic Minority: Psychoeducation App | Non-Hispanic: Usual Care | Racial / Ethnic Minority: Usual Care
Number analyzed (Participants) | 90 | 30 | 98 | 24 | 38 | 20
Participants
  Return Rate at Baseline | 89 | 29 | 98 | 24 | 38 | 19
  Return Rate at 3-month Follow up | 68 | 23 | 72 | 20 | 31 | 16
  Return Rate for both time points | 68 | 23 | 72 | 20 | 31 | 16

2. Primary Outcome: Feasibility of Fecal Sample Collection as Measured by Number of Participants Who Provide Fecal Samples
Description: as for outcome 1
Time Frame: Baseline and 3 month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Non-Hispanic White: HMP App | Racial / Ethnic Minority: HMP App | Non-Hispanic White: Psychoeducation App | Racial / Ethnic Minority: Psychoeducation App | Non-Hispanic: Usual Care | Racial / Ethnic Minority: Usual Care
Number analyzed (Participants) | 90 | 30 | 98 | 24 | 38 | 20
Participants
  Return Rate at Baseline | 90 | 30 | 98 | 24 | 37 | 20
  Return Rate at 3-month follow up | 69 | 24 | 72 | 20 | 30 | 17
  Return Rate both time points | 69 | 24 | 72 | 20 | 29 | 17

3. Secondary Outcome: Change in Microbiome Alpha Diversity: Species Richness
Description: Genetic analyses of the microbiome of the fecal sample (microorganism DNA, not that of the person) will be performed. Reported here are the observed (total number of distinct taxa) and calculated (Chao1 = N + S2 / (2 D), where N is the number of observed OTUs (Operational Taxonomic Units), S is the number of singleton OTUs, and D is the number of doublet OTUs) number of species represented in the sample. Chao1 is a species richness calculator that accounts for rare species.
Time Frame: Baseline and 3 month follow-up
Population: Samples were not received from all participants at all time points.
Measure: Mean (Standard Deviation); unit: species
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Number analyzed (Participants) | 91 | 92 | 46
species
  Observed at baseline: number analyzed (Participants) | 90 | 90 | 45
  Observed at baseline | 261.47 (143.66) | 271.59 (139.46) | 294.22 (130.35)
  Observed at 3-month follow up: number analyzed (Participants) | 91 | 87 | 46
  Observed at 3-month follow up | 257.34 (133.74) | 278.55 (143.96) | 295.67 (148.78)
  Calculated at baseline: number analyzed (Participants) | 90 | 90 | 45
  Calculated at baseline | 261.64 (143.82) | 271.84 (139.52) | 294.98 (130.68)
  Calculated at 3-month follow up: number analyzed (Participants) | 91 | 87 | 46
  Calculated at 3-month follow up | 257.57 (133.91) | 278.75 (144.07) | 295.96 (148.76)

4. Secondary Outcome: Change in Microbiome Alpha Diversity: Shannon Diversity Index (H')
Description: Genetic analyses of the microbiome of the fecal sample (microorganism DNA, not that of the person) will be performed. Shannon Diversity Index quantifies both the richness and the evenness of a community. It takes into account the number of taxa (richness) and their relative abundances (evenness). A higher Shannon index value indicates greater diversity, with both a high number of taxa and more even distribution of abundances among them. It is often used to assess the balance between species in a community. Typically ranges from 0-5 with higher numbers indicating increasing species diversity.
Time Frame: Baseline and 3 month follow-up
Population: Samples were not received from all participants at all time points.
Measure: Mean (Standard Deviation); unit: H' index
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Number analyzed (Participants) | 91 | 92 | 46
H' index
  diversity at baseline: number analyzed (Participants) | 90 | 90 | 45
  diversity at baseline | 4.28 (0.78) | 4.28 (0.74) | 4.35 (0.72)
  diversity at 3-month follow up: number analyzed (Participants) | 91 | 87 | 46
  diversity at 3-month follow up | 4.26 (0.76) | 4.33 (0.74) | 4.40 (0.73)

5. Secondary Outcome: Change in Microbiome Alpha Diversity: Inverse Simpson (1/D)
Description: Genetic analyses of the microbiome of the fecal sample (microorganism DNA, not that of the person) will be performed. Simpson is the probability that any two microbes are the same species, ranging from 0-1. Inverse Simpson (1 / Simpson) considers both richness and evenness. It places greater weight on the more abundant taxa. A higher inverse Simpson index suggests a more even distribution of taxa, with fewer dominant species. The inverse Simpson index is sensitive to the presence of dominant species and may emphasize diversity loss when one or a few species dominate the community.
Time Frame: Baseline and 3 month follow-up
Population: Samples were not received from all participants at all time points.
Measure: Mean (Standard Deviation); unit: 1/D index
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Number analyzed (Participants) | 91 | 92 | 46
1/D index
  Inverse Simpson at baseline: number analyzed (Participants) | 90 | 90 | 45
  Inverse Simpson at baseline | 62.75 (80.39) | 62.18 (77.51) | 60.73 (70.38)
  Inverse Simpson at 3-month follow up: number analyzed (Participants) | 91 | 87 | 46
  Inverse Simpson at 3-month follow up | 62.23 (78.81) | 64.07 (75.86) | 66.58 (75.16)

6. Secondary Outcome: Change in Microbiome Alpha Diversity: Pielou Evenness Index (J)
Description: Genetic analyses of the microbiome of the fecal sample (microorganism DNA, not that of the person) will be performed. Pielou Evenness Index measures how evenly the individuals are distributed across the taxa in a sample. It is calculated by dividing the Shannon diversity index by the maximum possible value of the Shannon index (which occurs when all taxa are equally abundant). The Pielou index ranges from 0 (no evenness, where one species dominates) to 1 (perfect evenness, where all species are equally abundant).
Time Frame: Baseline and 3 month follow-up
Population: Samples were not received from all participants at all time points.
Measure: Mean (Standard Deviation); unit: J index
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Number analyzed (Participants) | 91 | 92 | 46
J index
  Evenness Pielou baseline: number analyzed (Participants) | 90 | 90 | 45
  Evenness Pielou baseline | 0.78 (0.09) | 0.78 (0.09) | 0.78 (0.09)
  Evenness Pielou at 3-month follow up: number analyzed (Participants) | 91 | 87 | 46
  Evenness Pielou at 3-month follow up | 0.78 (0.09) | 0.79 (0.09) | 0.79 (0.09)

7. Secondary Outcome: Change in Microbiome Alpha Diversity: Simpson's Dominance Index (D)
Description: Genetic analyses of the microbiome of the fecal sample (microorganism DNA, not that of the person) will be performed. Simpson's Dominance Index measures the probability that two randomly selected individuals from a community belong to the same species (or taxon). It ranges from 0 to 1, where 0 indicates perfect diversity (no dominance of a single species) and values closer to 1 indicate that one or a few species dominate the community. A lower Simpson's dominance score suggests a more diverse community, while a higher score indicates a community dominated by a few taxa.
Time Frame: Baseline and 3 month follow-up
Population: Samples were not received from all participants at all time points.
Measure: Mean (Standard Deviation); unit: D index
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Number analyzed (Participants) | 91 | 92 | 46
D index
  Simpson's Dominance at baseline: number analyzed (Participants) | 90 | 90 | 45
  Simpson's Dominance at baseline | 0.03 (0.02) | 0.04 (0.03) | 0.03 (0.03)
  Simpson's Dominance at 3-month follow up: number analyzed (Participants) | 91 | 87 | 46
  Simpson's Dominance at 3-month follow up | 0.04 (0.02) | 0.03 (0.02) | 0.03 (0.02)

8. Secondary Outcome: Change in Inflammatory Biomarkers: C-reactive Protein
Description: Dried blood spot samples will be used to measure inflammatory cytokines (C-reactive protein (CRP) and interleukin-6 (IL-6)). Additionally mRNA assays will be used to detect and quantify inflammatory gene expression detect and monitor cellular immune responses. Analyses will focus on transcripts from ~200 genes known to be involved in the regulation of inflammation, and will consider key transcripts (e.g., IL-1beta, TNF-alpha) as well as summary measures reflecting the activity of transcriptional networks that coordinate inflammation (NF-kB, AP-1).
Time Frame: Baseline and 3 month follow-up
Population: only those who return their samples at both time points were included
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Number analyzed (Participants) | 91 | 92 | 47
mg/L
  baseline | 2.26 (4.17) | 2.40 (3.46) | 2.98 (4.67)
  3-month follow up: number analyzed (Participants) | 91 | 90 | 47
  3-month follow up | 2.62 (4.44) | 3.28 (5.30) | 3.10 (4.33)

9. Secondary Outcome: Change in Inflammatory Biomarkers: TNF-Alpha, IL-6, IL-10
Description: as for outcome 8
Time Frame: Baseline and 3 month follow-up
Population: only those who return their samples at both time points were included
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Number analyzed (Participants) | 91 | 92 | 47
pg/mL
  TNF-Alpha baseline: number analyzed (Participants) | 87 | 90 | 42
  TNF-Alpha baseline | 2.01 (5.58) | 1.54 (0.88) | 1.66 (0.67)
  TNF-Alpha 3-month follow up: number analyzed (Participants) | 88 | 90 | 45
  TNF-Alpha 3-month follow up | 1.73 (0.93) | 1.87 (0.84) | 1.98 (1.15)
  IL-6 baseline: number analyzed (Participants) | 87 | 90 | 42
  IL-6 baseline | 1.79 (13.20) | 0.26 (0.20) | 0.34 (0.39)
  IL-6 3-month follow up: number analyzed (Participants) | 88 | 90 | 45
  IL-6 3-month follow up | 0.98 (6.58) | 0.42 (0.83) | 0.98 (4.10)
  IL-10 baseline: number analyzed (Participants) | 87 | 90 | 42
  IL-10 baseline | 0.11 (0.12) | 0.10 (0.14) | 0.08 (0.07)
  IL-10 3-month follow up: number analyzed (Participants) | 88 | 90 | 45
  IL-10 3-month follow up | 0.13 (0.18) | 0.16 (0.26) | 0.11 (0.09)

10. Secondary Outcome: Change in Depression Symptoms Measured by Patient Health Questionnaire - 8 (PHQ-8) Score
Description: The PHQ-8 is an 8-item questionnaire where participants report how often in the past 2 weeks they were bothered by specific problems. It is scored on a 4-point Likert scale where 0 = not at all to 3 = nearly every day. The total possible range of scores is 0-24 where higher scores indicate more depressive symptoms.
Time Frame: Baseline, week 1, week 2, week 3, week 4 (of intervention period), and 3 month follow-up
Population: Survey participation dropped over time.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Number analyzed (Participants) | 120 | 122 | 58
score on a scale
  Baseline | 9.80 (4.74) | 9.91 (5.03) | 9.45 (4.57)
  Week 1: number analyzed (Participants) | 104 | 108 | 54
  Week 1 | 9.53 (5.02) | 9.30 (5.10) | 9.35 (4.70)
  Week 2: number analyzed (Participants) | 101 | 103 | 48
  Week 2 | 8.06 (4.87) | 8.35 (4.79) | 8.77 (4.49)
  Week 3: number analyzed (Participants) | 101 | 104 | 50
  Week 3 | 7.78 (4.68) | 7.88 (4.87) | 9.14 (4.43)
  Week 4: number analyzed (Participants) | 105 | 110 | 56
  Week 4 | 7.17 (4.89) | 7.44 (4.94) | 8.98 (4.38)
  3-month follow up: number analyzed (Participants) | 99 | 99 | 53
  3-month follow up | 6.78 (4.99) | 7.26 (5.13) | 7.81 (4.54)

11. Secondary Outcome: Change in Flourishing Measured by the Flourishing Index Score
Description: The Flourishing Index is a 10-item questionnaire where participants report their general level of flourishing (e.g., well-being, health, etc.). It is scored on a 0 to 10-point scale, with anchors varying across items. The total score ranges from 0 to 100 with higher scores indicating higher flourishing.
Time Frame: Baseline, week 1, week 2, week 3, week 4 (of intervention period), and 3 month follow-up
Population: Survey participation dropped over time.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Number analyzed (Participants) | 120 | 122 | 58
score on a scale
  Baseline | 55.61 (16.47) | 56.4 (16.75) | 57.14 (16.54)
  Week 1: number analyzed (Participants) | 104 | 109 | 53
  Week 1 | 56.31 (17.51) | 56.5 (14.36) | 57.62 (14.02)
  Week 2: number analyzed (Participants) | 101 | 103 | 48
  Week 2 | 60.39 (16.01) | 59.19 (14.92) | 57.26 (16.01)
  Week 3: number analyzed (Participants) | 101 | 104 | 50
  Week 3 | 62.11 (16.65) | 61.12 (15.53) | 57.65 (15.35)
  Week 4: number analyzed (Participants) | 105 | 110 | 56
  Week 4 | 63.64 (17.73) | 63.31 (15.75) | 59.10 (15.85)
  3-month follow up: number analyzed (Participants) | 99 | 99 | 53
  3-month follow up | 65.01 (18.34) | 63.47 (16.84) | 61.48 (14.09)

12. Other Pre Specified Outcome: Number of Participants With PHQ-8 Scores That Increased by 5 Points or More Compared to Baseline
Description: The PHQ-8 is an 8-item questionnaire where participants report how often in the past 2 weeks they were bothered by specific problems. Increase in scores indicates increase is depression symptoms.
Time Frame: Baseline, week 1, week 2, week 3, week 4 (of intervention period), and 3 month follow-up
Population: Survey participation dropped over time.
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Number analyzed (Participants) | 120 | 122 | 58
Participants
  baseline to Week 1: number analyzed (Participants) | 104 | 108 | 54
  baseline to Week 1 | 11 | 8 | 6
  baseline to Week 2: number analyzed (Participants) | 101 | 103 | 48
  baseline to Week 2 | 7 | 3 | 4
  baseline to Week 3: number analyzed (Participants) | 101 | 104 | 50
  baseline to Week 3 | 9 | 6 | 5
  baseline to Week 4: number analyzed (Participants) | 105 | 110 | 56
  baseline to Week 4 | 8 | 6 | 7
  baseline to 3-month follow up: number analyzed (Participants) | 99 | 99 | 53
  baseline to 3-month follow up | 8 | 6 | 3

ADVERSE EVENTS:
Time Frame: data collected up to 4 months on study
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/120 | 0/122 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/120 | 0/122 | 0/58
Other Adverse Events (participants affected / at risk) | 24/120 | 15/122 | 10/58
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Healthy Minds Program (HMP) App (N=120) | Psychoeducation App (N=122) | Usual Care (N=58)
Increased Symptoms of Depression (Psychiatric disorders) | 24 | 15 | 10 — Participants report how often in the past 2 weeks they were bothered by specific problems. Increase in scores PHQ-8 scores indicate increase is depression symptoms. This is the number of participants with increases of 5 points or more.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-16): https://cdn.clinicaltrials.gov/large-docs/01/NCT06213701/Prot_SAP_000.pdf